CLINICAL TRIAL: NCT00053391
Title: Vaccination Of HLA-A1 And/Or -A2+ Stage III or IV Melanoma Patients With Tumor Peptide - Loaded Autologous Dendritic Cells That Are Generated In The Absence Or Presence Of CD40 Ligand
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, PD Dr. med. univ. Beatrice Schuler-Thurner, Prinicipal Investigator Prof. Dr. Schuler Gerold, University Hospital Erlangen
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258491; ERLANGEN-1490; EU-20232
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — CD40 Ligand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: recombinant CD40-ligand
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with tumor proteins may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of vaccination with autologous dendritic cells pulsed with tumor and influenza antigen peptides treated with vs without ex vivo CD40-ligand, in terms of tumor-specific T-cell response, in patients with HLA-A1 and/or HLA-A2.1 positive stage III or IV melanoma.
* Determine the safety and tolerability of these vaccinations in these patients.
* Determine tumor response and recurrence rates in patients treated with these vaccinations.

OUTLINE: This is an open-label non-randomized study.

* Phase I: Patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMC). PBMC are cultured with sargramostim (GM-CSF) and interleukin-4 to generate dendritic cells (DCs) on day -9. DCs are pulsed separately with HLA-A1 and HLA-A2.1-restricted flu matrix peptides derived from melanoma-associated tumor antigens (MAGE-10.A2, Melan-A, MAGE-3, NY-ESO-1, gp100 antigen, and tyrosinase peptide). Half of the DCs are treated ex vivo with CD40-ligand. Patients receive the peptide-pulsed DC vaccinations subcutaneously (SC) on days 1, 14, 42, and 70 in the absence of disease progression.

Patients who show tumor response (at least stable disease) at day 98 progress to phase II of the study.

* Phase II: Patients undergo leukapheresis as in phase I on days 102, 352, and 688. Patients receive up to 6 additional booster vaccinations SC as in phase I on days 126, 184, 268, 356, 520, and 692.

Patients are followed for 10 years.

PROJECTED ACCRUAL: A total of 8-30 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV cutaneous malignant melanoma
* HLA-A1 and/or HLA-A2 expression by serologic HLA typing

  * HLA-A2.1 subtype must be confirmed by polymerase chain reaction on genomic DNA obtained from peripheral blood mononuclear cells
* No active CNS metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 4 months

Hematopoietic

* WBC greater than 2,500/mm^3
* Neutrophil count greater than 1,000/mm^3
* Lymphocyte count greater than 700/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin greater than 9 g/dL
* No bleeding disorders

Hepatic

* Bilirubin less than 2.0 mg/dL
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine less than 2.5 mg/dL

Cardiovascular

* No clinically significant heart disease

Pulmonary

* No clinically significant respiratory disease

Immunologic

* No active systemic infection
* No immunodeficiency disease

  * No evidence of HIV-1, HIV-2, or human T-cell lymphotropic virus-1
* No active autoimmune disease including (but not limited to):

  * Lupus erythematosus
  * Autoimmune thyroiditis or uveitis
  * Multiple sclerosis
  * Inflammatory bowel disease

Other

* Stable medical condition
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 month after study participation
* No organic brain syndrome or psychiatric illness that would preclude study compliance
* No other concurrent active malignancy
* No other concurrent serious illness that would preclude study treatment
* No contraindication to leukapheresis

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* No other concurrent immunotherapy

Chemotherapy

* More than 4 weeks since prior systemic chemotherapy (6 weeks for nitrosoureas)
* No concurrent chemotherapy

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to the spleen
* Concurrent palliative radiotherapy allowed

Surgery

* Recovered from prior surgery
* No prior splenectomy
* No prior organ allograft
* Concurrent surgery on selected metastases (e.g., because of pain or local complications such as compression) allowed

Other

* No other concurrent investigational drugs
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of vaccination with vs without ex vivo CD40-ligand in terms of tumor-specific T-cell response
Safety
Tolerability

SECONDARY OUTCOMES:
Tumor response
Recurrence rates

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Schuler, Study Chair — Dermatologische Klinik MIT Poliklinik-Universitaetsklinikum Erlangen
Locations (1):
- Dermatologische Klinik mit Poliklinik - Universitaetsklinikum Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Gross S, Erdmann M, Haendle I, Voland S, Berger T, Schultz E, Strasser E, Dankerl P, Janka R, Schliep S, Heinzerling L, Sotlar K, Coulie P, Schuler G, Schuler-Thurner B. Twelve-year survival and immune correlates in dendritic cell-vaccinated melanoma patients. JCI Insight. 2017 Apr 20;2(8):e91438. doi: 10.1172/jci.insight.91438. eCollection 2017 Apr 20. PMID 28422751